CLINICAL TRIAL: NCT04343079
Title: Intra-operative PET-CT: a Novel Approach to Determine Excision Margins in Lumpectomy Breast Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2017/0200
Record Dates: First submitted 2020-01-20; First posted 2020-04-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Female; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- braeast cancer (Experimental): breast cancer patients
  Interventions: Diagnostic Test: PET CT

INTERVENTIONS:
Diagnostic Test: PET CT — measurement of surgical margins during lumpectomy

SUMMARY:
Examination of the feasibility of intra-operative pet CT to detect surgical margins in breast conservative surgery to prevent re-excision.

ELIGIBILITY:
Inclusion Criteria:

* • female and 18 years of age or older

  * diagnosed with an early-stage (T1 or T2, and N0 or N1; according to the TNM-classification) invasive breast cancer
  * eligible for breast conserving surgery

Exclusion Criteria:

* • Pregnancy or lactation

  * Diabetes
  * Multifocal tumor disease
  * Diagnosis of inflammatory breast cancer
  * Appointment at the nuclear medicine department for 18F-FDG administration would result in a unacceptable delay of surgery
  * Subject has had exposure to ionizing radiation of more than 1 mSv in other research studies within the last 12 months
  * Subject has recently (<60 days) or is simultaneously participating in another clinical trial.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with breast cancer
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
investigate the ability of (micro)PET/CT to evaluate the excision margins and determine negativity of these margins, as compared to the gold standard of sectional histopathological evaluation. | 2 year
  study the feasibility of PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Oost Vlaanderen, Belgium

REFERENCES:
- [Derived] De Crem AS, Tummers P, Depypere H, Braems G, Salihi R, Vergauwen G, Cisternino G, Van de Vijver K, De Visschere P, De Man K, Van den Broeck B, Hendrickx S, Veldeman L, Monten C, Debacker JM, Denys H, Goker M. Breast cancer Intraoperative Margin Assessment using specimen PET-CT (BIMAP). NPJ Breast Cancer. 2025 Sep 26;11(1):101. doi: 10.1038/s41523-025-00818-8. PMID 41006264